CLINICAL TRIAL: NCT00065039
Title: Wise Mind: Environmental Approach for Obesity Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: YSMIND (completed)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise; Ethanol; Pharmaceutical Preparations; Tobacco Products

INTERVENTIONS:
Behavioral: Promotion of a healthy diet and physical activity
Behavioral: Avoidance of Alcohol, Drugs, and Tobacco

SUMMARY:
The study will be conducted in four Catholic schools with children enrolled in Grades 2 through 6. Girls and boys and children of all racial types are eligible for participation in the study. We anticipate that approximately 1,000 to 1200 children will volunteer for the study. We request enrollment of 1200 children. To participate, parents must grant written consent and the child must assent by signing a consent form that is attached. Two of the four schools that volunteer for participation in the study and are approved by the research team, will be randomly assigned to a health promotion program called "Wise Mind for Diet and Physical Activity. The other two schools will be randomly assigned to a program called "Wise Mind for Avoidance of Alcohol, Drugs, and Tobacco." Students will receive the program in the school that they attend. They will not be allowed to select one of the programs and will receive only one program, i.e., the program in their school. Both health promotion programs will last for two academic years. Each year, every child that is a research participant will be tested on two occasions, once during the first two months of school (Sept and Oct), and once during the last two months of school (March and April). Testing will not be conducted during May in order to avoid interference with school activities at the end of the academic year. All children (in all four schools) will have the same testing. The testing will involve confidential measurement of eating habits, food intake, physical activity habits, attitudes about alcohol, drugs, and tobacco, body weight and height, body fatness, body image, mood, and self-esteem. The measurement techniques that will be used for this measurement will include: questionnaires, weighing, measurement of height, and photography of foods before and after eating. All measurements will be confidential and will not be released to anyone that is not involved in the management of the study, including school personnel. The total time requirement for each testing period is expected to be approximately three hours, spread over four testing periods during a two-week period. The testing periods will be conducted in conjunction with school administrators and will not be scheduled to conflict with important school activities, classes, or academic tests. A Data and Safety Monitoring Board (DSMB) will be organized to provide oversight for the conduct of the study.

ELIGIBILITY:
* Must be a student in one of the four catholic schools in Baton Rouge that have elected to participate in the study.
* Must be in the second through sixth grade at the start of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Williamson DA, Han H, Johnson WD, Martin CK, Newton RL Jr. Modification of the school cafeteria environment can impact childhood nutrition. Results from the Wise Mind and LA Health studies. Appetite. 2013 Feb;61(1):77-84. doi: 10.1016/j.appet.2012.11.002. Epub 2012 Nov 12. PMID 23154216